CLINICAL TRIAL: NCT04137328
Title: Clinical Study on the Improvement of Diabetic Neuropathic Pain by Liraglutide
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Bin Lu, chief physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 358106
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Diabetic Neuropathic Pain
MeSH Terms: interventions — Liraglutide; Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- liraglutide group (Experimental): Mecobalamin tablets (0.5mg/day, oral) and liraglutide (0.6mg/day in the first week, if there is no obvious discomfort, 1.2mg/day in the second week, subcutaneous injection) were used for 3 months.
  Interventions: Drug: Liraglutide
- control group (Active Comparator): Take Mecobalamin (0.5mg/day, oral), add or adjust insulin (when basic insulin is preferred for those who do not use insulin, if insulin has been used, adjust the dose or program according to the condition, inject subcutaneously) for 3 months.
  Interventions: Drug: insulin

INTERVENTIONS:
Drug: Liraglutide — 0.6mg/day in the first week, if there is no obvious discomfort, 1.2mg/day in the second week, subcutaneous injection, lasting for 3 months
  Other Names: GLP-1RA
  Arms: liraglutide group
Drug: insulin — Add or adjust insulin (when basic insulin is preferred for those who do not use insulin, such as those who have already used insulin, adjust the dosage or program according to the condition, inject subcutaneously) for 3 months
  Arms: control group

SUMMARY:
Diabetic neuropathic pain is a common clinical manifestation of diabetic neuropathy, which seriously affects the quality of life of patients. The clinical treatment is limited and the curative effect is not good. In the previous animal studies, investigators found that the change of pain threshold in diabetic rats showed a staged change, and was significantly related to the change of brain microglia activity. It was confirmed that liraglutide could regulate the activation of microglia in vitro. Then investigators found that it could intervene diabetic neuropathic pain through the intervention of liraglutide in diabetic rats. In the early stage of clinical observation, the investigators also preliminarily observed that liraglutide can intervene diabetic neuropathic pain. At present, liraglutide is a commonly used hypoglycemic drug in clinic. Therefore, on the basis of previous studies, this study intends to select diabetic neuropathic pain patients whose blood sugar is not up to the standard, and give Mecobalamin to treat diabetic neuropathy. In addition, on the basis of the original hypoglycemic treatment, participants are randomly divided into one group to give liraglutide, one group to increase or adjust insulin, with similar blood glucose level. The improvement of diabetic neuropathic pain was observed. The aim of this study was to evaluate the safety and efficacy of liraglutide in improving diabetic neuropathic pain.

DETAILED DESCRIPTION:
1. Diabetic neuropathic pain seriously affects the quality of life, clinical problems are difficult, and new treatment methods are urgently needed.

Diabetic neuropathy is one of the most common complications of diabetes mellitus. The study of investigators shows that the prevalence rate of diabetic neuropathy diagnosed in downtown Shanghai is as high as 61.8%. The most common type of diabetic peripheral neuropathy is distal symmetric polyneuropathy, which is the main cause of diabetic neuropathic pain (DNP). Diabetic neuropathic pain can affect about one fifth of diabetic patients, which can lead to the decrease of daily activities, even the loss of work, severe depression, and quality of life. The pathogenesis of diabetic neuropathic pain is complex and not yet fully clear, so there is a lack of available and effective treatment. At present, the first-line clinical treatment drugs include pregabalin, duloxetine, amitriptyline, gabapentin and venlafaxine, etc., and these drugs sometimes relieve the symptoms of diabetic neuropathic pain not obvious, and have more side effects, which has become a difficult problem in clinical treatment. Therefore, it is urgent to explore effective drugs for diabetic neuropathic pain.

2. The clinical observation and animal study of the investigators show that the GLP-1 receptor agonist (liraglutide) can improve diabetic neuropathic pain.

1. Diabetic neuropathic pain is related to brain microglia. In the animal model of diabetes mellitus, investigators found the phenomenon of abnormal activation of microglia. Previous studies showed that the abnormal activation of microglia at the level of spinal cord was closely related to diabetic neuropathic pain, and microglia at the level of spinal cord played an important role in the transmission of pain. As the center of pain loop, the activity of microglia in cerebral cortex and thalamus is less related to diabetic neuropathic pain.

   Therefore, investigators used STZ induced diabetic neuropathy model of SD rats. Before STZ injection (0 week), at the 2nd, 4th, 6th and 12th week after STZ induced hyperglycemia. The investigators monitored the changes of body weight, blood glucose level and pain threshold of mechanical pain and thermal pain in rats. The investigators used [18F] dpa714 specific marker transfer protein TSPO to carry out PET / CT scan of brain to reflect microglia in each brain area. After PET / CT scan, EMG was used to evaluate the degree of peripheral nerve injury. The results showed that after STZ injection, compared with the control group, the blood glucose of STZ group increased gradually, and with the increase of blood glucose, the nerve conduction velocity of diabetic rats decreased gradually. Mechanical pain decreased significantly in 4-6 weeks, thermal pain threshold decreased significantly in 4 weeks, and mechanical pain and thermal pain sensitivity disappeared in 12 weeks. The results of PET / CT showed that in cortex, hippocampus, thalamus, hypothalamus and pituitary, dpa714 standard uptake value was significantly higher than other time points in the fourth week, and significantly higher than that in the control group. The correlation analysis indicated that the pain threshold of thermal pain was significantly related to the activity of microglia in thalamus and hypothalamus. Previous studies have shown that hyperglycemia can induce neuropathic pain. Thermal hyperalgesia occurs 4 weeks after hyperglycemia, while mechanical hyperalgesia occurs 4-6 weeks. PET / CT study showed that the activity of microglia in the brain of diabetic rats increased in the fourth week, and the activity of microglia was significantly related to the occurrence of heat pain. It has not been reported that the relationship between the activity of microglia and diabetic neuropathic pain was directly observed by PET / CT.
2. Liraglutide can regulate the activation of microglia Glucagon like peptide 1 (GLP-1) acts by binding to GLP-1 receptor, which is a G protein coupled receptor. A large number of studies have shown that GLP-1 receptor agonists can improve the activation of macrophages, microglia as macrophages in the brain, and GLP-1 receptor agonists can improve the activation of macrophages. However, few studies have shown that in vitro cultured astrocytes and microglia, GLP-1 analogues can change the morphology of glial cells, reduce IL-1 β and increase cAMP level at mRNA level.

   Therefore, liraglutide, the GLP-1 agonist, was selected as the intervention drug . BV2 microglia cell line was used as the following treatment methods: liraglutide was co cultured with LPS or high glucose, and liraglutide was added after LPS and high glucose induced activation. After treatment, the levels of IL-6 and TNF - α in the supernatant of the cells were observed. The results showed that liraglutide was added in advance before induction and activation. Or the level of IL-6 and TNF - α released by BV2 could be significantly reduced by using liraglutide. Therefore, liraglutide can regulate LPS and high glucose induced microglia activation.
3. Animal experiments show that liraglutide can improve diabetic neuropathic pain. On the basis of previous work, the investigators further studied the effect of liraglutide on diabetic neuropathic pain at the animal level. SD rats were divided into three groups: normal blood glucose group, normal saline control group and 200ug / kg / dliraglutide injection group. The latencies and thresholds of thermal and mechanical pain were monitored weekly. It was observed that for diabetic neuropathic pain rats, the peripheral injection of GLP-1 receptor agonist (liraglutide 200ug / kg / D) significantly increased the thermal pain threshold at 4 weeks, the mechanical pain threshold at 8 weeks, and the pain sensitivity disappeared at 12 weeks in both the normal saline control group and the liraglutide injection group.
4. Observation of clinical cases In clinical work, the investigators observed some obese patients with neuropathic pain in type 2 diabetes mellitus. In the process of using GLP-1 receptor agonist to control blood glucose, the symptoms of pain were also significantly improved. In addition, a clinical study showed that the use of sitagliptin (DPP-IV inhibitor, which can inhibit the degradation of GLP-1 in vivo) can also improve diabetic neuropathic pain. However, these observations and studies have significant limitations, not excluding the effect of blood glucose lowering itself in the population level, nor exploring the mechanism.

3. The clinical study of liraglutide in improving diabetic neuropathic pain has better clinical value.

The investigators found that liraglutide can improve the activation of microglia, and it can significantly alleviate diabetic neuropathic pain at the animal level and clinical cases. The systematic study of liraglutide used to improve neuropathic pain in diabetic patients has not been reported, and this subject has better clinical value.

Therefore, considering the hypoglycemic effect of liraglutide on the basis of previous studies, the investigators plan to select diabetic neuropathic pain patients whose blood sugar is not up to standard in this study, and give Mecobalamin (one of the commonly used drugs recommended in the guidelines for prevention and treatment of diabetes mellitus to treat neuropathy). At the same time, on the basis of the original hypoglycemic treatment, participants were randomly divided into one group to be given liraglutide and the other group to be increased/adjusted insulin. After 3 months, the improvement of diabetic neuropathic pain in the two groups under the condition of similar blood glucose level were observed. The purpose of this study was to evaluate the safety and efficacy of liraglutide in improving diabetic neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 and ≤ 80; The patients were diagnosed as type 2 diabetic neuropathic pain, and the score of pain digital scoring method was more than 3 points; 7-9% of glycosylated hemoglobin had poor blood glucose control.

Exclusion Criteria:

Non diabetic neuropathic pain; BMI < 20kg / m2; There are serious primary diseases such as cardiovascular, liver, kidney and hematopoietic system; In the past 1 month, there were acute complications such as diabetic ketoacidosis, lactic acidosis and hyperosmotic coma; Over the past five years, there have been alcoholics and / or psychoactive substances, drug abusers and addicts; Pregnant or lactating women; Unwillingness to cooperate or various factors affecting compliance; Psychopaths; Those who have participated in other clinical projects in the past 1 month.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-30 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Numerical pain scale (NRS) | 3 months
  The number of 0-10 represents the degree of pain of the patient, 0 is no pain, 10 is extreme pain. How to write: circle the number that describes the most severe pain in the last 24 hours.

SECONDARY OUTCOMES:
Neurological symptom score (NSS) / neurological deficit score (NDS) | 3 months
  Clinical diagnosis criteria of diabetic neuropathy: NDS score ≥ 6 points or NDS score 3-5 points with NSS score ≥ 5 points
Examination of nerve conduction function | 3 months
  The examination of nerve conduction function was completed by professional doctors of EMG room using EMG evoked potential instrument. During the test, the patient was relaxed and lying in a quiet room, and the skin temperature was maintained at 32 ℃ ~ 33 ℃. Motor nerve examination includes: measurement of motor nerve conduction velocity, compound muscle action potential amplitude and distal latency of median nerve, ulnar nerve, common peroneal nerve and tibial nerve; sensory nerve examination includes: measurement of sensory nerve conduction velocity and action potential amplitude of median nerve, ulnar nerve, superficial peroneal nerve and sural nerve.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Lu, doctor, Study Director — Huashan Hospital

IPD SHARING:
Plan to Share IPD: No
we have no plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Background] Jeffcoate WJ, Vileikyte L, Boyko EJ, Armstrong DG, Boulton AJM. Current Challenges and Opportunities in the Prevention and Management of Diabetic Foot Ulcers. Diabetes Care. 2018 Apr;41(4):645-652. doi: 10.2337/dc17-1836. PMID 29559450
- [Background] Lu B, Yang Z, Wang M, Yang Z, Gong W, Yang Y, Wen J, Zhang Z, Zhao N, Zhu X, Hu R. High prevalence of diabetic neuropathy in population-based patients diagnosed with type 2 diabetes in the Shanghai downtown. Diabetes Res Clin Pract. 2010 Jun;88(3):289-94. doi: 10.1016/j.diabres.2010.02.002. Epub 2010 Mar 31. PMID 20359765
- [Background] Kanera IM, van Laake-Geelen CCM, Ruijgrok JM, Goossens MEJB, de Jong JR, Verbunt JA, Geerts M, Smeets RJEM, Kindermans HPJ. Living with painful diabetic neuropathy: insights from focus groups into fears and coping strategies. Psychol Health. 2019 Jan;34(1):84-105. doi: 10.1080/08870446.2018.1518526. Epub 2018 Oct 15. PMID 30320508
- [Background] Tsuda M. Microglia in the spinal cord and neuropathic pain. J Diabetes Investig. 2016 Jan;7(1):17-26. doi: 10.1111/jdi.12379. Epub 2015 Jun 23. PMID 26813032
- [Background] Inoue K, Tsuda M. Microglia in neuropathic pain: cellular and molecular mechanisms and therapeutic potential. Nat Rev Neurosci. 2018 Mar;19(3):138-152. doi: 10.1038/nrn.2018.2. Epub 2018 Feb 8. PMID 29416128
- [Background] Hirano T, Mori Y. Anti-atherogenic and anti-inflammatory properties of glucagon-like peptide-1, glucose-dependent insulinotropic polypepide, and dipeptidyl peptidase-4 inhibitors in experimental animals. J Diabetes Investig. 2016 Apr;7 Suppl 1(Suppl 1):80-6. doi: 10.1111/jdi.12446. Epub 2016 Mar 31. PMID 27186361
- [Background] Bruen R, Curley S, Kajani S, Crean D, O'Reilly ME, Lucitt MB, Godson CG, McGillicuddy FC, Belton O. Liraglutide dictates macrophage phenotype in apolipoprotein E null mice during early atherosclerosis. Cardiovasc Diabetol. 2017 Nov 6;16(1):143. doi: 10.1186/s12933-017-0626-3. PMID 29110715
- [Background] Vinue A, Navarro J, Herrero-Cervera A, Garcia-Cubas M, Andres-Blasco I, Martinez-Hervas S, Real JT, Ascaso JF, Gonzalez-Navarro H. The GLP-1 analogue lixisenatide decreases atherosclerosis in insulin-resistant mice by modulating macrophage phenotype. Diabetologia. 2017 Sep;60(9):1801-1812. doi: 10.1007/s00125-017-4330-3. Epub 2017 Jun 12. PMID 28608285
- [Background] Lee CH, Jeon SJ, Cho KS, Moon E, Sapkota A, Jun HS, Ryu JH, Choi JW. Activation of Glucagon-Like Peptide-1 Receptor Promotes Neuroprotection in Experimental Autoimmune Encephalomyelitis by Reducing Neuroinflammatory Responses. Mol Neurobiol. 2018 Apr;55(4):3007-3020. doi: 10.1007/s12035-017-0550-2. Epub 2017 Apr 29. PMID 28456941
- [Background] Barros JI, Fechine FV, Montenegro Junior RM, Vale OC, Fernandes VO, Souza MH, Cunha GH, Moraes MO, d'Alva CB, Moraes ME. Effect of treatment with sitagliptin on somatosensory-evoked potentials and metabolic control in patients with type 2 diabetes mellitus. Arq Bras Endocrinol Metabol. 2014 Jun;58(4):369-76. doi: 10.1590/0004-2730000002914. PMID 24936731